CLINICAL TRIAL: NCT06636097
Title: Effect of the Intaglio Surface of Full-arch Implant-supported on Marginal Bone Level: A Cross-sectional Study
Brief Title: Intaglio Surface of Full-arch Implant Supported Prosthesis
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Andrea Ravida, Assistant Professor, University of Pittsburgh
Other Study IDs: STUDY23100028
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Peri-Implantitis
Keywords: Peri-implantitis; Marginal Bone Level; Dental Implants; Full-arch Prosthesis; Hybrid prosthesis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Bacterial collection will be collected from the implant sulcus and from the abutments of the prosthesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients Rehabilitated with full-arch implant-supported prosthesis: All patients that are rehabilitated with full-arch implant-supported prosthesis
  Interventions: Device: Full arch

INTERVENTIONS:
Device: Full arch — design

SUMMARY:
The purpose of the study is to determine if there is an association between the intaglio shape of full-arch implant-supported prosthesis and marginal bone level around implants. The intaglio shape can be present as concave or convex and, depending on that, it can lead to more plaque accumulation on the fitting surface of the prosthesis.

Null Hypothesis (H0): Full-arch implant supported prosthesis with an increased depth of the intaglio shape demonstrate similar marginal bone levels as prosthesis with a reduced depth of the intaglio surface.

Alternative Hypothesis (H1): Full-arch implant supported prosthesis with an increased depth of the intaglio shape demonstrate increased/reduced marginal bone levels compared to prosthesis with a reduced depth of the intaglio surface.

DETAILED DESCRIPTION:
The investigators will review dental records from the university and call eligible individuals for an appointment. During the research visit, the investigators will take new x-rays for marginal bone level assessment and a digital scan of the prosthesis to assess the shape of the intaglio. Also, remove the prosthesis, perform clinical measurements and collect plaque samples from the prosthesis and the implant sulcus. then, implants and prosthesis will be cleaned and placed in position.

The study will have only one appointment where every measurement will be assessed in this visit.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old;
* Rehabilitated with a full-arch screw-retained supported prosthesis in the maxilla, in function for at least 1 year;
* Good overall health (ASA I or ASA II).

Exclusion Criteria:

* Individuals with motricity problems who cannot clean the prosthesis;
* Patients treated or maintained in centers outside the University of Pittsburgh;
* Incomplete dental records;
* Misfit at the prosthesis-implant interface;
* Cemented prosthesis;
* Individuals rehabilitated with over dentures;
* Individuals with uncontrolled chronic diseases or immunocompromised;
* Pregnant Patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients treated with a full-arch implant-supported prothesis from the University of Pittsburgh will be screened for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the depth of the shape of the intaglio surface of full-arch and its association with increased marginal bone level. | The measurements will be assessed during the unique visit of the patient in the study.
  After the prosthesis is scanned, and evaluation of the 3D file of the prosthesis will occur. A virtual line will be traced between the Buccal to the Palatal/Lingual flange of the prosthesis. In the middle point of this line, a perpendicular line will be traced in direction of the fitting surface of the prosthesis, intaglio, and this distance will be measured in mm.

SECONDARY OUTCOMES:
Probing Depth of the implants | The measurements will be assessed during the unique visit of the patient in the study.
  Using a periodontal probe we will register Probing Depth in 6 sites per implant. All measures will be in mm.
Bleeding on Probing of the implants | The measurements will be assessed during the unique visit of the patient in the study.
  Using a periodontal probe we will register Bleeding in 6 sites using the bleeding indexes modified for dental implants.
Modified Plaque Index | The measurements will be assessed during the unique visit of the patient in the study.
  Plaque accumulation will be evaluated using the modified plaque index adapted for dental implants.
Marginal Recession | The measurements will be assessed during the unique visit of the patient in the study.
  The distance, in mm, between the implant platform and the mucosal margin.
Suppuration | The measurements will be assessed during the unique visit of the patient in the study.
  Assessed by the presence/absence of suppuration after gentle probing of the implants.
Keratinized mucosa width | The measurements will be assessed during the unique visit of the patient in the study.
  Measured from the mucosal marginal level of the implants to the mucogingival junction. The band of keratinized mucosa will be characterized as narrow < 2mm and wide > 2mm.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ravida, DDS, MS, PhD, Principal Investigator — Program Director of the Periodontics and Implant Dentistry Department
Locations (1):
- University of Pittsburgh, School of Dental Medicine, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Mombelli A, van Oosten MA, Schurch E Jr, Land NP. The microbiota associated with successful or failing osseointegrated titanium implants. Oral Microbiol Immunol. 1987 Dec;2(4):145-51. doi: 10.1111/j.1399-302x.1987.tb00298.x. No abstract available. PMID 3507627
- [Result] Araujo MG, Lindhe J. Peri-implant health. J Periodontol. 2018 Jun;89 Suppl 1:S249-S256. doi: 10.1002/JPER.16-0424. PMID 29926949